CLINICAL TRIAL: NCT01914952
Title: Alternate Dosing Strategies for Beta-hydroxy-beta-methylbutyrate (HMB) Supplementation: Effect on Plasma HMB Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MTI2013-CS02
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Focus of the Study is to Examine Plasma HMB Levels After Oral HMB Supplementation
Keywords: CaHMB; HMB free acid; HMB
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CaHMB Capsule (Active Comparator)
  Interventions: Dietary Supplement: CaHMB capsule
- HMB free acid gelcap (Active Comparator)
  Interventions: Dietary Supplement: HMB free acid gelcap
- HMB free acid in water (Active Comparator)
  Interventions: Dietary Supplement: HMB free acid mixed in water
- CaHMB powder in water (Active Comparator)
  Interventions: Dietary Supplement: CaHMB in water
- HMB free acid (oral not in gelcap or water) (Active Comparator)
  Interventions: Dietary Supplement: HMB free acid

INTERVENTIONS:
Dietary Supplement: CaHMB capsule — 1.0 gram of CaHMB powder in a gelatin capsule
  Arms: CaHMB Capsule
Dietary Supplement: HMB free acid gelcap — 0.8 g HMB free acid is a soft gel capsule
  Arms: HMB free acid gelcap
Dietary Supplement: HMB free acid mixed in water — 0.8 g HMB free acid in water
  Arms: HMB free acid in water
Dietary Supplement: CaHMB in water — 1.0 g CaHMB powder mixed in water
  Arms: CaHMB powder in water
Dietary Supplement: HMB free acid — 0.8 g HMB free acid
  Arms: HMB free acid (oral not in gelcap or water)

SUMMARY:
The purpose of this study is to examine the rise in plasma Beta-hydroxy-beta-methylbutyrate (HMB) after the dietary supplement has been administered in different forms. Prior studies have indicated that form of administration affects bioavailability of the HMB supplement. Therefore the current study will examine the bioavailability of a single dose of HMB given as:

* 1.0g CaHMB in gelatin capsule
* 0.8 g HMB free acid in a gelcap
* 0.8 g HMB free acid in water
* 1.0 g CaHMB in water
* 0.8 g HMB free acid

The randomized study will be a crossover design and each study subject will undergo the experimental protocol for each of the supplementation forms. Because of the different administration forms, the study will be an open label study. Briefly, the fasted participants will report to the laboratory in the morning. After an initial blood sample is taken, the dose of HMB will be administered. Blood will then be samples at 2, 5, 10, 15, 25, 35, 45, 60, 90, 120, 180, 360, 720, and 1440 min post administration. A 24 h complete urine collection will also be performed. Participants will be given a light sack lunch 4 h after administration of the dosage and will remain at the laboratory through the 360 min sampling. Participants will then be allowed to leave the laboratory and return for the 720 min sampling after which the participants can eat an normal evening meal. Participants will return to the laboratory fasted the next morning for the final sample. A minimum 48 h washout period will be required before the next dosage form is administered and the process repeated.

ELIGIBILITY:
Inclusion Criteria:

* Must not be taking amino acid, protein, or HMB supplements; Must not be pregnant; Must not be breastfeeding

Exclusion Criteria:

* Currently taking amino acid, protein, or HMB supplements; Currently pregnant; Currently breastfeeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Plasma HMB Level | Plasma samples collected at 0, 2, 5, 10, 15, 25, 35, 45, 60, 90, 120, 180, 360, 720, and 1440 min after treatment administration

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States